CLINICAL TRIAL: NCT00002443
Title: Twelve-Month Study in HIV-1 Seropositive Retroviral-Naive Patients to Compare the Safety and Efficacy of MK-639 and Zidovudine (AZT) Administered Concomitantly to MK-639 Alone and Zidovudine (AZT) Alone
Brief Title: The Safety and Effectiveness of MK-639 and Zidovudine, Used Alone and Together, in HIV-Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 246B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Zidovudine

SUMMARY:
To compare the effects on CD4 counts and safety of MK-639 (indinavir, IDV) and AZT administered concomitantly to MK-639 alone and AZT alone in HIV-1 seropositive patients.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 3 groups for 12 months of treatment. Group 1 receives MK-639 plus AZT. Group 2 receives MK-639 alone. Group 3 receives AZT alone. Safety and tolerability are assessed by the incidence of clinical and laboratory adverse experiences. Blood and urine samples are collected for safety assessment and to determine CD4 cell counts and serum viral RNA levels. If therapy with MK-639 alone or with AZT is found to be generally safe and clinically efficacious, patients who have completed the study will have the opportunity to continue in an extension study protocol on a treatment regimen including MK-639.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* Average CD4 count between 50 and 500 cells/mm3 based on 2 separate pre-study determinations at least 1 week apart.

Note:

* Patients with known hemophilia may be enrolled at the discretion of the investigator.

Prior Medication:

Excluded:

* Any protease inhibitor.
* Significant prior use (greater than 2 weeks) of nucleoside analogues.
* Chronic therapy for an active opportunistic infection. (Allowed:
* Prophylaxis with aerosolized pentamidine, trimethoprim/sulfamethoxazole, dapsone, topical antifungals, and isoniazid).
* Investigational agents or immunomodulators within 30 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Acute hepatitis.
* Lymphoma.
* Visceral Kaposi's sarcoma.
* Invasive cervical cancer.
* Active infection.

Concurrent Medication:

Excluded:

Anticipated immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780
Dates: Study Completion 1996-01